CLINICAL TRIAL: NCT02363530
Title: Influence of 2% HPMC Used During Cataract Surgery for Intraoperative Corneal Optical Clarity and Post-operation Xerophthalmia.
Brief Title: Corneal Protect Used During Cataract Surgery
Acronym: CPUDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Wangshu Yu, Eye Center of the Second Affiliated Hospital, School of Medicine, Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Corneal Protect
Record Dates: First submitted 2015-02-05; First posted 2015-02-16 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Cataract
Keywords: cataract surgery; cornea protect; xerophthalmia; Corneal clarity
MeSH Terms: conditions — Cataract; Xerophthalmia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPMC group (Experimental): Patients use the intervention Hydroxypropyl ethylcellulose (HPMC) 2% gel during the cataract surgery.
  Interventions: Device: Hydroxypropyl ethylcellulose (HPMC) 2% gel
- BSS group (Placebo Comparator): Patients use balanced salt solution (BSS) during the cataract surgery.
  Interventions: Device: BSS

INTERVENTIONS:
Device: Hydroxypropyl ethylcellulose (HPMC) 2% gel — We use the hydroxypropyl ethylcellulose (HPMC) 2% gel instead of the traditional balanced salt solution during the cataract surgery.
  Other Names: Cornea Protect
  Arms: HPMC group
Device: BSS — Balanced Salt Solution including normal saline and glucose
  Other Names: Balanced Salt Solution
  Arms: BSS group

SUMMARY:
This randomized controlled subject- and examiner-masked study comprised patients scheduled for cataract surgery.The patients will be randomly assigned to receive either balanced salt solution（BSS）or hydroxypropyl methylcellulose（HPMC）2% gel （Cornea Protect）.Each subject should undertake examination including - rupture time (TBUT), height of the river of tears, fluorescence staining, Schirmer Ⅰ test, ocular surface disease index (OSDI) and self-conscious symptom assessment questionnaire for assessment.

DETAILED DESCRIPTION:
This randomized controlled subject- and examiner-masked study comprised patients scheduled for cataract surgery.Over 100 patients will be randomly assigned to receive either balanced salt solution（BSS）or hydroxypropyl methylcellulose（HPMC）2% gel （Cornea Protect）.Each subject will accept 5 times assessments:the day before surgery, surgery day , the day after surgery,a week after surgery and a month after surgery.Each time a subject should undertake examination including - rupture time (TBUT), height of the river of tears, fluorescence staining, Schirmer Ⅰ test, ocular surface disease index (OSDI) and self-conscious symptom assessment questionnaire et.al.The purpose is to evaluate the effect of Cornea Protect to maintain intraoperative clarity and to prevent the postoperative xerophthalmia.

ELIGIBILITY:
Inclusion Criteria:

* with cataracts;
* aged 40 to 85 years old, gender not limited;
* plans to accept PHACO and intraocular lens(IOL)implantation surgery
* the lens nucleus hardness level is less than 3 ;
* signed informed consent.

Exclusion Criteria:

* allergic to any of the drugs or device in this study ；
* existence of other infectious diseases or allergic conjunctivitis.
* the eye had been chemical burned or thermal burned
* diagnosed as Stevens Johnson syndrome or eye-pemphigoid.
* diagnosed with glaucoma or high intraocular pressure;
* existence of eyelid and lacrimal duct disease;
* received any eye surgery in 3 months;
* wearing corneal contact lens;
* history suggests there are serious heart, lung, liver or renal function disorder;
* pregnancy or lactation women;
* Other conditions considered not appropriate by the investigators.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline dry eye condition at 1 month | an expected average of a month after the surgery
  Dry eye condition includes tear break up time (TBUT), height of the river of tears,Schirmer Ⅰ test,ocular surface disease index (OSDI) and self-conscious symptom assessment questionnaire.
Intraoperative corneal clarity | during the surgery
  record the times of using HPMC or BSS during the surgery to maintain the intraoperative corneal clarity and how long it lasts.
change from baseline corneal damage at 1 month | an expected average of a month after the surgery
  Corneal damage evaluated by fluorescence staining of cornea

SECONDARY OUTCOMES:
Inflammation | an expected average of a month after the surgery
  Inflammation evaluated by Anterior chamber scintillation
change from baseline dry eye condition at 1 week | an expected average of a week after the surgery
  Dry eye condition includes tear break up time (TBUT), height of the river of tears,Schirmer Ⅰ test,ocular surface disease index (OSDI) and self-conscious symptom assessment questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Yao, PhD, Principal Investigator — Eye Center of the Second Affiliated Hospital of Zhejiang University
Locations (1):
- Eye Center of the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Chen YA, Hirnschall N, Findl O. Comparison of corneal wetting properties of viscous eye lubricant and balanced salt solution to maintain optical clarity during cataract surgery. J Cataract Refract Surg. 2011 Oct;37(10):1806-8. doi: 10.1016/j.jcrs.2011.07.001. Epub 2011 Jul 22. PMID 21782381